CLINICAL TRIAL: NCT05108350
Title: A Single-centre, Parallel-cohort, Randomized, Open-label, Two-period, Cross-over, Bioequivalence Study of the Fixed Dose Combination of HR20033 Relative to Co-administration of the Individual Components in Two Cohorts of Healthy Chinese Subjects in the Fed State
Brief Title: A Study to Assess the Bioequivalence of Fixed Dose Combination of HR20033 Relative to Co-administration of the Individual Components in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR20033-101
Record Dates: First submitted 2021-11-03; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: There will be two independent cohorts of subjects who will each receive two treatments (high dose strength and low dose strength), and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability. In each cohort approximately 40 healthy subjects will be randomized to receive treatment with IP to complete at least 36 evaluable subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HR20033 FDC 5/500 mg (Experimental)
  Interventions: Drug: T1: FDC 5/500 mg; R1+R: SHR3824 5 mg + Metformin 500 mg XR
- SHR3824 5mg + Metformin 500 mg XR (Experimental)
  Interventions: Drug: T1: FDC 5/500 mg; R1+R: SHR3824 5 mg + Metformin 500 mg XR
- HR20033 FDC 5/1000 mg (Experimental)
  Interventions: Drug: T2: FDC 5/1000 mg; R2+R: SHR3824 5 mg + two Metformin 500 mg XR
- SHR3824 5 mg + Metformin 1000 mg XR (Experimental)
  Interventions: Drug: T2: FDC 5/1000 mg; R2+R: SHR3824 5 mg + two Metformin 500 mg XR

INTERVENTIONS:
Drug: T1: FDC 5/500 mg; R1+R: SHR3824 5 mg + Metformin 500 mg XR — SHR3824 5 mg + Metformin 500 mg XR In cohort 1 (low dose strength), subjects will receive treatment T1 followed by 7 days washout and then receive treatment R1+R.
  Arms: HR20033 FDC 5/500 mg
Drug: T1: FDC 5/500 mg; R1+R: SHR3824 5 mg + Metformin 500 mg XR — SHR3824 5 mg + Metformin 500 mg XR In cohort 1 (low dose strength), subjects will receive treatment R1+R followed by 7 days washout and then receive treatment T1.
  Arms: SHR3824 5mg + Metformin 500 mg XR
Drug: T2: FDC 5/1000 mg; R2+R: SHR3824 5 mg + two Metformin 500 mg XR — SHR3824 5 mg + Metformin 1000 mg XR In cohort 2 (high dose strength), subjects will receive treatment T2 followed by 7 days washout and then receive treatment R2+R.
  Arms: HR20033 FDC 5/1000 mg
Drug: T2: FDC 5/1000 mg; R2+R: SHR3824 5 mg + two Metformin 500 mg XR — SHR3824 5 mg + Metformin 1000 mg XR In cohort 2 (high dose strength), subjects will receive treatment R2+R followed by 7 days washout and then receive treatment T2.
  Arms: SHR3824 5 mg + Metformin 1000 mg XR

SUMMARY:
The trial is to assess the bioequivalence between HR20033 FDC tablet and co-administration of SHR3824 tablets and metformin XR tablets.

The primary objective is to evaluate bioequivalence of SHR3824 and Metformin in healthy Chinese subjects in the fed state.

The secondary objective is to evaluate the safety of HR20033 FDC tablet in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process, and possible adverse reactions of the trial;
2. Must be able to communicate with the investigator, understand and comply with all study requirements;
3. Subject (include their fere) must have not pregnancy plan from 2 weeks prior to dose administration to 6 months after last dose administration and must use effective form of birth control;
4. Male or female subjects aged 18 to 50 (including 18 and 50);
5. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 18 and <28 kg/m2. BMI = weight (kg)/[height (m)]2;
6. No clinically significant deviation from normal in medical history, vital signs, physical examination.

Exclusion Criteria:

1. Regular smoker within 3 months prior to study drug administration, or quitting smoking less than 30 days until screening;
2. History of allergy to test drugs, allergic constitution (multiple drug and food allergies);
3. A history of alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); those who have abstained from alcohol have not quit for 30 days at the time of screening;
4. Donate blood or lose a lot of blood (>450mL) within three months before screening;
5. Take any drugs that alter liver enzyme activity 28 days before screening;
6. Take any prescription drugs, over-the-counter drugs, any vitamin products or herbal medicines within 14 days before screening;
7. Those who have taken a special diet (including pitaya, mango, grapefruit, etc.) or exercised vigorously within 2 weeks before screening, or other factors that affect drug absorption, distribution, metabolism, and excretion;
8. Combine the following inhibitors or inducers of CYP3A4, P-gp or Bcrp, such as itraconazole, ketoconazole or dronedarone;
9. Significant changes in diet or exercise habits recently;
10. Have taken the research drug or participated in the drug clinical trial within three months before taking the research drug;
11. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption;
12. Suffer from any diseases that increase the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
13. Subjects who cannot tolerate standard meals (two boiled eggs, a slice of buttered bacon toast, a box of fried potato chips, a cup of whole milk);
14. Abnormal ECG has clinical significance;
15. Female subjects are breastfeeding or have a positive serum pregnancy result during the screening period or the test;
16. Clinical laboratory tests have clinically significant abnormalities, or other clinical findings in the 12 months before screening show clinical significance for the following diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune , Mental or cardiovascular disease);
17. Viral hepatitis (including hepatitis B and C), AIDS antibody, and Treponema pallidum antibody screening are positive (for those with Treponema pallidum antibody positive, additional RPR testing is required);
18. Acute illness or concomitant medication from the screening stage to the study medication;
19. Ingested chocolate, any caffeine-rich or xanthine-rich food or drink 48 hours before taking the study drug;
20. Have taken any alcohol-containing products or a positive alcohol breath test within 48 hours before taking the study medication;
21. Those who have a positive urine drug screen or have a history of drug abuse in the past five years;
22. Have been exposed to metformin and/or SGLT2 inhibitor drugs such as dapagliflozin, empagliflozin, canagliflozin, and empagliflozin within 1 month before administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-09 (Estimated); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Cmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: AUC0-t | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: AUC0-inf (if applicable) | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8

SECONDARY OUTCOMES:
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Tmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: Vz/F | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: CL/F | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin in the fasted and fed state: t1/2 | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Tmax | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Ctrough | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
Pharmacokinetics parameters of SHR3824 and Metformin after single and multiple dose: Racc etc | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8
The incidence and severity of adverse events/serious adverse events | Based on pre-dose, 0.5-72 hours post-dose sampling times on Day 1 and Day 8

IPD SHARING:
Plan to Share IPD: Undecided